CLINICAL TRIAL: NCT05714410
Title: Evaluation of Changes in Bowel Movement Frequency Following the Consumption of Partially Hydrolyzed Guar Gum (PHGG) in Adults with Constipation As Compared to Placebo (Typhoon 2)
Brief Title: Evaluation of Changes in Bowel Movement Frequency Following the Consumption of PHGG Compared to Placebo
Acronym: TYPHOON-02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 22.08.CLI
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: Constipation - Functional

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PHGG fiber (Active Comparator): Partially Hydrolyzed Guar Gum (PHGG) in powder formulation, is to be consumed orally adding water or juice. One serving per day.
  Interventions: Dietary Supplement: PHGG
- Placebo Maltodextrin (Placebo Comparator): Maltodextrin in powder formulation is to be consumed orally adding water or juice. One serving per day.
  Interventions: Dietary Supplement: PHGG

INTERVENTIONS:
Dietary Supplement: PHGG — PHGG

SUMMARY:
Evaluation of Changes in Bowel Movement Frequency Following the Consumption of Partially Hydrolyzed Guar Gum (PHGG) in Adults With Constipation as Compared to Placebo (Typhoon 2)

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18-75.
2. Adapted Rome IV Criteria of functional constipation* or IBSconstipation** for a minimum of 3 months

   *1-2 SBM/week and at least 1 of the following at least 30% of the time:
   1. Bristol stool scale 1-2
   2. Straining
   3. Sense of incomplete evacuation
   4. Sense of stool blockage
   5. Need of digital maneuvers

      * Subjects with IBS-C: the above constipation criteria + abdominal pain are allowed.
3. Ability to understand the participant information sheet and instructions, and able to provide informed consent.
4. Access to a suitable smartphone device (Android or iOS) with ability to download and complete the study e-Diary daily for the duration of the trial.

Exclusion Criteria:

1. Pregnant women or breastfeeding.
2. Organic chronic gastrointestinal disease or complication (such as, but not limited to, Inflammatory Bowel Disease, Microscopic colitis, Eosinophilic gastroenteritis, Radiation-related enterocolitis, Coeliac disease).
3. Subjects with a diagnosed food allergy or hypersensitive to any of the components of the study product.
4. Subjects with chronic diarrhea.
5. Active peptic ulcer.
6. Major gastrointestinal or colonic surgery (such as, gastric bypass or any other obesity or metabolic interventions including endoscopic procedures or devices, any gastro-intestinal or colonic resection); cholecystectomy and appendectomy are allowed.
7. Neurologic or other clinically significant comorbid diseases that may affect gastrointestinal function, such as multiple sclerosis, spinal cord injury or Hirschsprung disease.
8. Illness that may preclude the participant's ability to complete the study or that may confound the study outcomes (e.g. bowel cancer, prostate cancer, terminal illness, severe cardiovascular disease, chronic renal failure or eating disorders) or any other serious illness resulting in >2 weeks inability to work in the 3 months before the study start.
9. Participants with clinically significant (as per physician judgement) co-morbid illnesses such as cardiovascular, endocrine (e.g. hypothyroidism, diabetes), renal, or other chronicdisease (e.g. reduced mobility or increased fragility).
10. Active alcohol, drug, or medication abuse (as per clinician judgement).
11. Self-reported symptoms suggestive of pelvic organ prolapse as per clinician judgement, such as feeling of pressure or fullness in the pelvic area, intra vaginal discomfort, painful intercourse, and urinary problems.
12. Moderate or severe active local anorectal problems such as recurrent anal fissures, frequent bleeding, large prolapsing hemorrhoids.
13. Any clinically relevant abnormalities detected during the physical examination or any alarm features in the medical history such as sudden unintentional weight loss (>10% in 3 months), frequent rectal bleeding not caused by anal fissures or hemorrhoids, recent change in bowel habit (<3 months), severe abdominal pain and stool positive for occult blood.
14. Regular (i.e. daily or weekly) use of PHGG within 6 months of screening.
15. Participation in another study with any investigational product within 6 months of randomization for drug study and within 2 months of randomization for a nutritional study.
16. Investigator believes that the participant is physically or mentally unfit to participate in the trial.
17. Participants currently of childbearing potential, but not using an effective method of contraception, as determined by the investigator.
18. Any participant who is an employee of the study site or an Atlantia Clinical Trials employee or their close family member or a member of their household.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Change in Spontaneous Bowel Movements | 6 weeks
  Change in mean weekly frequency of Spontaneous Bowel Movements (SBM) as measured by the daily bowel diary from baseline to end of treatment period. Frequency will be defined as the mean weekly number of SBM during the 2-week run-in period prior to V0, for baseline, and during the final 2 weeks of the intervention period, for end of treatment.

SECONDARY OUTCOMES:
Change in frequency of Complete Spontaneous Bowel Movements | 6 weeks
  Change in mean weekly frequency of Complete Spontaneous Bowel Movements (CSBM) as measured by the daily bowel diary, from baseline to the end of treatment period.
Change in stool consistency | 6 weeks
  Change in stool consistency as measured by the Bristol stool scale, from baseline to end of intervention. The minimum and maximum values are 1 to 7. The extremes scores mean worse outcome. The middle or the scale mean the better outcome.
Change in constipation related symptoms | 6 weeks
  Change in constipation related symptoms from baseline to end of intervention as measured by the Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire. The minimum and maximum values are 1 to 48. The higher score means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Muckley, FRCPI, Principal Investigator — Altantia Food Clinical Trial
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No